CLINICAL TRIAL: NCT02713750
Title: Optimization of Reproductive Health Care for Female Adolescents Living With HIV (Reproductive Health in HIV-infected Female Adolescents)
Brief Title: RH and Adolescents
Status: Completed | Type: Observational
Sponsor: The HIV Netherlands Australia Thailand Research Collaboration (Other)
Collaborators: amfAR, The Foundation for AIDS Research (Other); ViiV Healthcare (Industry)
Responsible Party: Sponsor
Other Study IDs: HIV-NAT 176
Record Dates: First submitted 2016-03-09; First posted 2016-03-21 (Estimated); Last update posted 2016-03-21 (Estimated); Status verified 2016-03

CONDITIONS: Reproductive Health
Keywords: Combined Oral Contraceptives; Highly Active Antiretroviral Therapy; Hormonal Contraception; Human Immunodeficiency Virus; Intrauterine Device; Pharmacokinetic; Sexually Transmitted Diseases; Reproductive Health
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome; Sexually Transmitted Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- HIV female adolescents: sexually active, HIV-infected female adolescents, 12-24 years old who are aware of their HIV status
  Interventions: Other: reversible contraceptive methods

INTERVENTIONS:
Other: reversible contraceptive methods — 1. Consistent male condom use only
  2. Consistent female condom use only
  3. Hormonal contraception, combined oral contraceptive pills and male/female condom
  4. Hormonal contraception, progestin only depot medroxyprogesterone acetate (DMPA) injectable and male/female condom
  5. Hormonal contraception , progestin only hormonal implant and male/female condom
  6. Intrauterine device and male/female condom

SUMMARY:
This study will create a model of reproductive health services for HIV-positive female adolescents in Asia.

DETAILED DESCRIPTION:
For the implementation of risk reduction interventions, it is equally important to provide specific knowledge and continuous counseling on different preventive options. A perfect preventive method, which provides highly reliable dual protection both from unintended pregnancies and from HIV/STDs with no side effects and which is completely accepted, is not available. Many authors consider that the most effective way to achieve dual protection is the simultaneous use of two contraceptive methods, one of which is a barrier method such as the male or female condom, and the other a highly effective contraceptive method, such as hormonal contraception (HC), intrauterine device (IUD) or sterilization. This is called dual contraception. Therefore this project will focus on specific reproductive service delivery for these groups of patients. As the age group is very young, the investigators will use in the study only reversible highly effective methods of contraception - HC, combined or progestin only, and an IUD - and condoms. For example, HC for HIV-positive women has been studied extensively in the last two decades, yet there are still no definitive answers regarding key issues - HIV disease progression, genital tract HIV shedding and infectivity, pharmacokinetic (PK) interactions between hormones and ARVs, and therefore a possibility for compromise of contraceptive effect and/or ARV failure, and last but not least, metabolic outcomes. Data on the effect of hormonal contraception on HIV disease progression is still inconclusive. Unfortunately there is only a limited number of studies in this field, with very small sample sizes and in most cases outside "real life" conditions.

There are three substudies:

1. Pharmacokinetic interactions between the sex steroid hormones and the protease inhibitors in HIV-positive Thai female adolescents
2. Assessment of premenstrual syndrome in HIV-positive adolescents
3. Metabolic changes in HIV + female adolescents on ART with hormonal contraception

ELIGIBILITY:
Inclusion Criteria:

* Female 12 to 24 years of age
* HIV-positive status
* HIV-disclosed before screening visit
* Having had first menstrual cycle (menarche)
* Sexually active
* Willing to participate in the study and signed informed consent form, including signed inform consent by caretaker for subjects <18 years of age

Exclusion Criteria:

* Being pregnant at the time of screening visit
* Mental or physical conditions that may limit informed participation in the study
* Having active AIDS or opportunistic infections

Non-eligible subjects to use hormonal contraception:

* Thrombosis or history of it
* Family history of thrombosis
* Hypertension (for combined oral contraceptives)
* Hyperlipidemia (toxicity grade >3)
* Diabetes mellitus with vascular involvement
* Presence or history of liver hepatic disease
* Malignant disease of genital organs and breast
* Undiagnosed vaginal bleeding
* Lactation
* Hypersensitivity to steroid hormones

Eligible subjects to use intrauterine device:

* In case of HAART, last CD4 count > 200 cells/mm3 no more than 6 months prior to the screening
* If without HAART, last CD4 count >350 cells/mm3 no more than 6 months prior to the screening
* Normal cervical Pap smear in the last 6 months/in the day of IUD insertion

Non-eligible subjects to use intrauterine device:

* Having an active infection of the vagina or cervix
* Having pelvic inflammatory disease (PID) or have a recent history of PID
* Having a bleeding disorder or taking anticoagulants
* Having abnormalities of the uterus
* Having a uterine infection after childbirth or a septic abortion
* Having uterine bleeding of unknown origin
* Having an allergy to copper

Ages: 12 Years to 24 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: 100 sexually active, HIV-infected female adolescents, 12-24 years old. All subjects should know their HIV status.
Sampling Method: Non-Probability Sample
Enrollment: 77 (Actual)
Dates: Start 2013-03; Primary Completion 2015-11 (Actual); Study Completion 2015-11 (Actual)

PRIMARY OUTCOMES:
number of participants who use any of the proposed contraceptive methods | 18 months
number of participants who adhere to the use of the proposed contraceptive mthods | 18 months

CONTACTS AND LOCATIONS:
Locations (4):
- Thailand (4):
  - HIV-NAT, Thai Red Cross AIDS Research Centre, Bangkok
  - Phramongkutklao Hospital of The Royal Thai Army, Bangkok
  - Srinagarind Hospital, Khon Kaen University, Khon Kaen
  - Phachomklao Hospital, Phetchaburi

REFERENCES:
- [Result] Kancheva Landolt N, Bunupuradah T, Achalapong J, Kosalaraksa P, Petdachai W, Ngampiyaskul C, Auchieng C, Ananworanich J, Boonyanurak P. Premenstrual Disorders Among Perinatally HIV-Infected Adolescents. J Acquir Immune Defic Syndr. 2015 Dec 1;70(4):e150-3. doi: 10.1097/QAI.0000000000000762. No abstract available. PMID 26181814